CLINICAL TRIAL: NCT01911351
Title: High Concentration Continuous Flow Nitrous Oxide Use for Procedural-induced Pain or Anxiety During Pediatric Minor Procedures
Brief Title: Nitrous Oxide Use in Minor Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2013-296
Record Dates: First submitted 2013-07-24; First posted 2013-07-30 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-02

CONDITIONS: Laceration; Abscess
Keywords: nitrous oxide; pediatric pain and anxiety
MeSH Terms: conditions — Lacerations; Abscess; Anxiety Disorders | interventions — Nitrous Oxide; Entonox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard management (No Intervention): Patients randomized to this arm will receive standard management alone for their minor procedure.
- Nitrous Oxide (Experimental): Patients randomized to this arm will receive nitrous oxide plus standard management for their minor procedure.
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous Oxide — Patients randomized to the intervention arm will receive nitrous oxide plus standard management for their minor procedure.
  Other Names: nitronox
  Arms: Nitrous Oxide

SUMMARY:
Title:

High-concentration continuous flow nitrous oxide use for procedural-induced pain or anxiety during pediatric minor procedures.

Objective: To assess whether the use of high-concentration continuous flow nitrous oxide in addition to standard management increases the comfort level in pediatric patients undergoing minor procedures compared to standard management alone.

DETAILED DESCRIPTION:
Title:

High-concentration continuous flow nitrous oxide use for procedural-induced pain or anxiety during pediatric minor procedures

Brief Summary:

Background: Over the past 10 years pediatric emergency departments (PED) throughout the country have adopted the concept of an "ouchless" PED, using both pharmacologic and non-pharmacologic methods to achieve this goal. There are a number of minor procedures performed routinely in a PED. Despite our interest in an "ouchless" PED, many of these procedures are performed without full attention to patient comfort. Some procedures, such as laceration repair, require local anesthesia, while others, such as intravenous catheter placement, are usually performed without local anesthesia. All of these minor procedures, however, are ones in which the risk of parenteral procedural sedation outweighs the benefit.

Due to the awareness of trying to create as pain-free an experience as possible, the use of high-concentration nitrous oxide (>50%) in the pediatric outpatient setting has grown and is used in PEDs throughout the country. Nitrous oxide is a colorless, non-narcotic, analgesic gas. Its efficacy and safety have been well documented in anesthesia, pediatric and dental literature. Over the last 30 years, nitrous oxide has been incorporated in the outpatient pediatric setting for procedural analgesia. At Jacobi Medical Center (JMC), nitrous oxide has been successfully used for children undergoing a variety of minor procedures in the PED.

Several studies have been published on the use of nitrous oxide in decreasing pain and anxiety in the pediatric emergency setting; however, previous studies using high concentration nitrous oxide have been either observational, have focused on a narrow age range, a single procedure type or procedures associated with moderate to severe pain, such as fracture reduction.

This investigation, unlike previous studies, will include a wider age range of children, as well as a variety of painful or anxiety provoking minor procedures commonly performed in the PED. We are choosing to include a variety of pre-defined minor procedures, rather than a single procedure, in order to assess the feasibility and benefit of nitrous oxide for the many minor procedures performed routinely on a daily basis in a pediatric emergency department. It will allow us to quantify our rate of effectiveness in decreasing pain and/or anxiety with the use of high concentration (>50%) nitrous oxide and to expand the use of nitrous oxide if shown to be superior to standard management in the reduction of procedural pain and anxiety.

Objective: To assess whether the use of high-concentration continuous flow nitrous oxide in addition to standard management increases the comfort level in pediatric patients undergoing minor procedures compared to standard management alone.

Methods: This will be a prospective randomized controlled trial conducted in the JMC PED. Children 3-12 years of age presenting to the PED, who require a minor procedure will be assessed for eligibility. Minor procedures will be defined as any procedure in which the standard management may involve providing local anesthetic and/or holding the child in order to successfully accomplish the procedure. These are not procedures in which the patient would receive parenteral analgesics, anxiolytics or anesthetics, because they are minimally painful and do not warrant the potential risks associated with parenteral anesthesia. Examples of minor procedures include simple incision and drainage of an abscess, intravenous catheter placement, urinary catheter placement, paronychia incision, foreign body removal and simple laceration repair. A local anesthetic such as injectable lidocaine or a topical anesthetic such as Eutectic Mixture of Local Anesthetics (EMLA) is frequently used and their use will be at the discretion of the provider performing the procedure. The doses of the topical anesthetics used are uniform. The decision of whether topical anesthesia will be used will be made by the provider before group randomization of the patient. Exclusion criteria include patients with medical conditions in which nitrous oxide is contraindicated, who are unable to communicate reliable levels of pain or who have low-to-no anxiety levels demonstrable by a validated anxiety scale, scored in the examining room by a research assistant after the procedure is described by the provider. After obtaining parental consent/child assent, patients will be randomized using a random number table to group 1 (nitrous oxide plus standard management) or group 2 (standard management alone). Because younger children especially experience significant anxiety before and during procedures, which can negatively affect the success of the procedure, we will use block randomization by groups of 6 for two separate age groups in order to ensure equal representation in both groups. These groups will be divided into preschool age (3 years to <6 years) and school age (>6 years- 12 years) children. Patients in the nitrous oxide group will receive nitrous oxide up to 70% concentration using a nitrous oxide protocol previously developed for use in the PED (attached), along with standard management (+/- local anesthetic, +/- holding the child) as determined by the provider prior to randomization. Patients in Group 2 will receive standard management alone (+/-local anesthetic, +/- holding the child).

Data Collection:

Data collection occurs at three time points: pre- procedure, intra-procedure and post-procedure. The pre-procedural data collection will include: 1) a pain score using a standard number scale ranging from 0-10 for children >6 years or 10-point Wong-Baker faces pain scale for children < 6 years measured at the time of triage by the triage nurse and 2) demographics including age, gender, procedure type, adjunctive pain medication (including the use of local anesthesia) and anxiety score using the Modified Yale Preoperative Anxiety Scale (M-YPAS) performed by a research assistant (medical student or college student who will be trained in data collection) in the treatment room after the provider has described the procedure to the patient and parent. Intra-procedural data collection will include: comfort score measured on the Face, Legs, Activity, Cry, Consolability (FLACC) Pain Scale and anxiety score measured on the M-YPAS. The FLACC Scale is a 10 point scoring system with 10 indicating the highest level of pain. Both scoring scales are validated scales of pain (FLACC) and anxiety (M-YPAS). The FLACC score and the M-YPAS score will be documented by a research assistant (medical student or college student who will be trained in data collection). The post-procedure data collection will include: mask tolerance, level of holding the child required in order to complete the procedure, length of procedure, highest nitrous oxide concentration used, patient recovery time back-to-baseline, adverse events, and independent rating of the success of the procedure by both the provider performing the procedure and the provider administering the nitrous oxide. At the end of the visit, a research assistant blinded to the patient's group assignment will document the parent's satisfaction with the encounter.

Outcomes:

The primary outcome will be the FLACC Pain Scale score measured intra-procedure. Secondary outcomes will be the M-YPAS Anxiety Score, length of the procedure, parent satisfaction score, and provider rating of success of the procedure. To assess inter-relator reliability, a second provider will complete the provider survey for 75% of the participants.

Sample Size:

Based on a pre-study sample of children undergoing minor procedures, the mean FLAAC Pain Scale score was 7.25/10. We determined that a 25% difference in the mean FLACC scores between the two groups would be clinically relevant. In various published articles a clinical significant change in pain score was noted with the use of nitrous oxide between 20% and 40%. At an alpha of .05 and a power of 80%, we estimate a sample size of 42 patients in each arm (21 patients in each of the two age ranges per arm).

Statistics:

Data will be collected and analyzed using Statistical Package for the Social Sciences (SPSS) version 19 with the FLACC Pain Scale being the primary outcome measure. The mean FLACC score will be compared between the two groups. Ordinal variables will be analyzed using the Mann-Whitney -U test and categorical values using the Chi Square test. Associations between the intra-procedure FLACC Pain Scale score with patient age (preschool and school age), pre-procedural pain and pre-procedural anxiety scores will be analyzed using Spearman correlation and the Chi Square test. The kappa statistic will be used to assess agreement between the two providers' rating of the success of the procedure. Since the randomization is stratified and the sample size calculation is based on stratified analysis, we will analyze both groups separately to test this hypothesis. An interim review of the data will be done effectiveness of the treatment. Any adverse events will be reported by the principal investigator in writing to the The Committee on Clinical Investigations (CCI) and the institutional review board (IRB).

Additional Response:

Although lack of blinding may be seen as a potential weakness concerning objectivity of the main outcome, we are intentionally not blinding the study in order to mimic PED practice. Our goal is to determine whether nitrous oxide will benefit the child in terms of reducing pain and/or anxiety during a minor procedure. The method of delivery, however, may be in itself noxious to some children (face mask). Introducing this aspect to the standard arm may unduly increase the FLACC Pain Scale score in this group. Additionally, in the sense that we may be introducing a noxious stimulus without any possibility of benefit seems unethical.

In both arms, the administration of local anesthetic and/or the degree to which a child is held in order to perform the procedure will be at the discretion of the treating physician. The practice, however, for a specific minor procedure is similar between all providers. For example, a child receiving sutures will have a topical anesthetic placed at triage and then injectable lidocaine administered at the time of the suturing. The doses for topical anesthetics are uniform and the decision by the provider whether to use topical anesthesia will be made before group randomization. In order for our data to be clinically meaningful, we again want to mimic PED practice. The details of all aspects of adjuvant care, such as local anesthetic use and holding a child, will be documented.

Risks:

The adverse effects of nitrous oxide occur very infrequently. However, in the literature, the following adverse effects have been described: vomiting, oxygen desaturation, dizziness, euphoria, abdominal pain and hallucinations.

Benefits:

The subjects may or may not experience a decreased pain and anxiety level, potential for shorter procedure time due to compliance, and increased parent/child satisfaction. A positive procedural experience may reduce long-term procedural traumatic distress.

ELIGIBILITY:
Inclusion Criteria:

* Minor Procedure
* Age 3 - 12 years

Exclusion Criteria:

* Behavioral Disorders
* Anxiety Score <10

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Cunningham, MD, Principal Investigator — Jacobi Medical Center - NYHHC
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Management | Nitrous Oxide
Started | 39 | 43
Completed | 39 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Management | Nitrous Oxide | Total
Number analyzed (Participants) | 39 | 43 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 43 | 82
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 5 [4 to 8] | 6 [4 to 9] | 5 [4 to 8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 25 | 26 | 51
Region of Enrollment [Number; unit: participants]
  United States | 39 | 43 | 82

OUTCOME MEASURES:

1. Primary Outcome: FLACC Pain Scale
Description: The primary outcome will be the FLACC (Face, Legs, Activity, Cry, Consolability) Pain scale measured intra-procedure. The scale measures facial expression, movement of legs, general activity, presence and quality of cry and the need and ability to be consoled. Scoring for each category ranges from 0 (no response to pain) to 2 (maximum response to pain). The scores are totaled and a total score ranging from 0-10 is reported.
Time Frame: peak pain during procedure approximately 2-5 minutes into the procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Management | Nitrous Oxide
Number analyzed (Participants) | 39 | 43
units on a scale | 8 [5 to 10] | 2 [0 to 5]

2. Secondary Outcome: M-YPAS Anxiety Scale
Description: Secondary outcome will be the Modified YALE Preoperative Anxiety Scale, measured pre-procedure, and intra-procedure. This is a validated scale measuring anxiety by assessment of Activity, Vocalization, Emotional Expressivity, State of Arousal and Use of Parents. All categories have a maximum score of 4 except for Vocalization with a maximum score of 6. The scores within each category are totaled and a total anxiety score is reported ranging from 5 (no anxiety) to 22 (highest level of anxiety).
Time Frame: measured pre-procedure at time provider explains procedure to the patient, and during procedure at peak pain time approximately 2-5 minutes into the procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Management | Nitrous Oxide
Number analyzed (Participants) | 39 | 43
units on a scale
  Preprocedural YPAS score | 14 [12 to 18] | 14 [12 to 18.5]
  intraprocedural YPAS score | 20 [15 to 22] | 10 [5 to 15]

3. Other Pre Specified Outcome: Length of the Procedure
Description: Another outcome measure is to compare the change in length of the procedure with or without nitrous oxide intervention.
Time Frame: measure time duration of each procedure, average 5-15 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Standard Management | Nitrous Oxide
Number analyzed (Participants) | 39 | 43
minutes | 11 [5 to 20] | 11 [5 to 16]

4. Other Pre Specified Outcome: Percentage of Parents Who Reported That Their Child Was Comfortable During the Procedure
Description: A parental survey was collected post-procedure regarding the overall comfort of the child during the procedure. Other questions included whether the procedure was successfully completed, if the procedure went better than expected, was the parent pleased with the medications used and whether the child tolerated the procedure. Answers were Strongly Agree, Agree, Neutral, Disagree and Strongly Disagree. We chose the question that asked whether the child was comfortable during the procedure as it was most relevant. The categories "Strongly Agree" and "Agree" were combined in both groups.
Time Frame: measured at the end of each procedure, approximately 10 minutes after the procedure is completed
Population: In the Standard Management arm, 38/39 parents completed the survey
Measure: Number; unit: percentage of participants
Arm/Group | Standard Management | Nitrous Oxide
Number analyzed (Participants) | 38 | 43
percentage of participants | 71 | 91

5. Other Pre Specified Outcome: Percentage of Providers Who Rated the Procedure as Being Successful
Description: Survey collection of rating of success of the procedure by one provider. Answers were Strongly Agree, Agree, Neutral, Disagree and Strongly Disagree. The first two categories were combined.
Time Frame: measured at the end of each procedure, approximately 10 minutes after the completion of the procedure
Measure: Number; unit: percentage of participants
Arm/Group | Standard Management | Nitrous Oxide
Number analyzed (Participants) | 39 | 43
percentage of participants | 70 | 91
Statistical Analysis 1: Comparison: Standard Management vs Nitrous Oxide; A kappa statistic was performed for 75% of the group to assess inter-rater agreement of the perception of the success of the procedure; Test type: Superiority or Other; p < 0.001, Chi-squared — A priori threshold for statistical significance: p< or = 0.05; kappa statistic = 0.88

ADVERSE EVENTS:
Description: Continuous real time observation
Arm/Group | Standard Management | Nitrous Oxide
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/43
Other Adverse Events (participants affected / at risk) | 0/39 | 3/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Management (N=39) | Nitrous Oxide (N=43)
hallucinations (Injury, poisoning and procedural complications) | 0 | 1
emesis (Injury, poisoning and procedural complications) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes